CLINICAL TRIAL: NCT05288504
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of AVTX-002 for the Treatment of Poorly Controlled Non-Eosinophilic Asthma
Brief Title: A Study to Evaluate the Safety and Efficacy of AVTX-002 for the Treatment of Poorly Controlled Non-Eosinophilic Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVTX-002-NEA-201
Record Dates: First submitted 2022-03-08; First posted 2022-03-21 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Non-Eosinophilic Asthma
Keywords: Non-Eosinophilic Asthma; AVTX-002

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AVTX-002 (Experimental): Approximately 40 subjects will receive AVTX-002 at a dose of 600 mg three times during the study.
  Interventions: Drug: AVTX-002
- Placebo (Placebo Comparator): Approximately 40 subjects will receive placebo sourced as normal saline three times during the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AVTX-002 — Dose of 600 mg administered subcutaneously three times during the study.
  Other Names: CERC-002, AEVI-002, MDGN-002
  Arms: AVTX-002
Drug: Placebo — Placebo sourced as normal saline administered subcutaneously three times during the study.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of AVTX-002 compared with placebo in patients with poorly controlled non-eosinophilic asthma (NEA).

ELIGIBILITY:
Inclusion Criteria:

* Documented non-eosinophilic asthma diagnosis (<300 eosinophils/μL).
* Symptoms consistent with a diagnosis of asthma that is poorly controlled as determined by an ACQ score ≥ 1.5.
* Poorly controlled asthma despite the use of a Long-Acting Beta-Agonists and Inhaled Corticosteroid for at least 3 consecutive months immediately prior to screening.
* Subjects must have had at least one asthma exacerbation in the last 24 months.

Exclusion Criteria:

* Pulmonary disease other than asthma.
* Currently on biologic therapy. Previous biologic therapy is permitted with adequate washout (12 weeks or 5 half-lives, whichever is longer).
* Use of systemic immunosuppressants within the last 6 months.
* Use of systemic corticosteroids within 6 weeks prior to Screening or use of antibiotics within 4 weeks prior to Screening.
* Subject has alanine aminotransferase (ALT)/ aspartate aminotransferase (AST) >5 upper limit of normal (ULN) and/or serum creatinine concentration >1.5 mg/dL.
* Subject has hemoglobin ≤10 g/dL, neutrophils ≤1,500/μl, and/or platelets ≤75,000/μl.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Garry Neil, MD, Study Director — Avalo Therapeutics, Inc.
Locations (24):
- United States (24):
  - Tucson Neuroscience Research - M3, Wake Research, Tucson, Arizona
  - Center For Clinical Trials of Sacramento, Sacramento, California
  - Allergy and Asthma Medical Group of the Bay Area, Walnut Creek, California
  - Center For Clinical Trials of San Gabriel, West Covina, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - National Jewish Health, Denver, Colorado
  - Helix Biomedics, LLC, Boynton Beach, Florida
  - Suncoast Research Group LLC, Miami, Florida
  - Suncoast Research Associates LLC, Miami, Florida
  - Pro-Care Research Center, Corp., Miami Gardens, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - ASHA Clinical Research-Munster, LLC, Hammond, Indiana
  - Family Allergy and Asthma Research Institute, Louisville, Kentucky
  - Continental Clinical Solutions, LLC, Towson, Maryland
  - Pulmonary Research Institute of Southeast Michigan, Farmington Hills, Michigan
  - Midwest Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, Lincoln, Nebraska
  - OK Clinical Research, Edmond, Oklahoma
  - Affinity Health, Nashville, Tennessee
  - Amarillo Center For Clinical Research, Amarillo, Texas
  - South Texas Medical Research Institute, Inc, Boerne, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Meridian Clinical Research, Portsmouth, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AVTX-002 | Placebo
Started | 45 | 46
Safety Analysis Set | 45 | 45
Full Analysis Set | 45 | 45
Per Protocol Analysis Set | 43 | 41
PK Analysis Set | 45 | 0
Completed | 36 | 32
Not Completed | 9 | 14

BASELINE CHARACTERISTICS:
Population: Randomized Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | AVTX-002 | Placebo | Total
Number analyzed (Participants) | 45 | 46 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (14.60) | 47.6 (15.99) | 46.6 (15.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 17 | 14 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 12 | 26
  Not Hispanic or Latino | 31 | 34 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 10 | 27
  White | 28 | 35 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 46 | 91
Weight [Mean (Standard Deviation); unit: kg] | 95.60 (23.661) | 87.94 (21.343) | 91.73 (22.722)
Height [Mean (Standard Deviation); unit: cm] | 168.41 (9.900) | 167.69 (10.865) | 168.04 (10.347)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 33.95 (8.917) | 31.20 (6.329) | 32.56 (7.798)
Screening eosinophil level [Count of Participants; unit: Participants]
  < 150 eosinophils per micro liter | 24 | 25 | 49
  >= 150 eosinophils per micro liter | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: The Ability of AVTX-002 to Improve Asthma Control in Subjects With Poorly Controlled Non-eosinophilic Asthma (NEA) Based on the Percentage of Patients Who Experience Asthma Related Events.
Description: Percentage of patients who experience any of the following asthma related events:
  * ≥6 additional reliever puffs of Short-Acting Beta-Agonist (compared to baseline) in a 24-hour period on 2 consecutive days or,
  * increase in inhaled corticosteroid dose ≥4 times than the dose at baseline or,
  * a decrease in peak flow of 30% or more (compared to baseline) on 2 consecutive days of treatment, or
  * an asthma exacerbation requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days, or
  * a hospitalization or emergency room visit because of an asthma exacerbation
Time Frame: Through Week 14
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 45 | 45
Participants | 12 | 14

2. Secondary Outcome: Change From Baseline to Week 14 in Forced Expiratory Volume in 1 Second (FEV1[Liters]).
Description: The FEV1 is the volume of air that can be forcibly exhaled from the lungs in the first second, measured in liters by a spirometer.
Time Frame: Through Week 14
Population: Full Analysis Set with all subjects with baseline and Week 14 data available.
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 42 | 42
Liter | -0.149 (0.309) | -0.203 (0.405)

3. Secondary Outcome: Time to Asthma Exacerbation.
Description: Time to event will be measured in days using the first day of the event to denote the day of the overall asthma related event occurrence.
Time Frame: Through Week 14
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 45 | 45
days
  Time to first asthma related event or time to censoring | 84.9 (28.03) | 78.1 (30.58)
  Time to first asthma related event - Subjects with an asthma related event: number analyzed (Participants) | 12 | 14
  Time to first asthma related event - Subjects with an asthma related event | 52.1 (31.83) | 42.6 (26.69)

4. Secondary Outcome: Change From Baseline to Week 14 in Fractional Exhaled Nitric Oxide (FeNO).
Description: A FeNO test measures the levels of nitric oxide during exhalation. A FeNO test will be done by breathing into a tube attached to a hand-held monitor.
Time Frame: Through Week 14
Population: Full Analysis Set with all subjects with baseline and Week 14 data available.
Measure: Mean (Standard Deviation); unit: Parts per billion
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 42 | 42
Parts per billion | 6.1 (15.54) | 3.8 (27.64)

5. Secondary Outcome: Change From Baseline to Week 14 in Asthma Control Questionnaire (ACQ).
Description: This is a simple questionnaire to measure the adequacy of asthma control and change in asthma control. ACQ has a multidimensional construct assessing symptoms (5 items, self-administered), rescue bronchodilator use (1 item, self-administered), and FEV1 (1 item, completed by study staff). Scores range between 0 (totally controlled) and 6 (severely uncontrolled).
Time Frame: Through Week 14
Population: Full Analysis Set with all subjects with baseline and Week 14 data available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 42 | 42
score on a scale | -0.22 (1.077) | -0.34 (0.999)

6. Secondary Outcome: Change From Baseline to Week 14 in Standardized Asthma Quality of Life Questionnaire for 12 Years and Older (AQLQ(S)+12).
Description: The AQLQ(S)+12 is a modified version of the standardized AQLQ and includes 32 questions in 4 domains (symptoms, activity limitation, emotional function, and environmental stimuli). Subjects will be asked to recall their experiences during the previous 2 weeks and score each of the questions on a 7-point scale, where 7=not at all limited and 1=totally limited. The overall score of the AQLQ +12 will be derived as the average of the 32 questions; thus, the total score ranges from 1 (indicates "total impairment") to 7 (indicates "no impairment").
Time Frame: Through Week 14
Population: Full Analysis Set with all subjects with baseline and Week 14 data available.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 42 | 42
score on a scale | 0.18 (1.423) | 0.49 (1.162)

7. Secondary Outcome: Change From Baseline to Week 14 in Asthma Symptom Diary Score.
Description: The Asthma Symptom Diary is a 6-item daily measure of asthma symptom severity that assesses three core categories of asthma symptoms: breathing symptoms (difficulty breathing; wheezing; shortness of breath), chest symptoms (chest tightness; chest pain), and cough. Subjects are required to rate the 6 symptoms at their worst each day using an 11-point numeric rating scale ranging from 0 ('None') to 10 ('As bad as you can imagine'). The Asthma Symptom Diary score is the sum of the 6 individual symptom scores (the range is from 0-60, where a higher score indicates more severe symptoms) reported as a weekly average.
Time Frame: Through Week 14
Population: Full Analysis Set with all subjects with baseline and Week 14 data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 35 | 28
units on a scale | -0.15 (1.469) | -0.39 (1.318)

8. Secondary Outcome: Change From Baseline to Week 14 in European Quality of Life - 5 Dimension 5 Level Questionnaire in Visual Analogue Scale Score (EQ VAS).
Description: The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ VAS. The EQ VAS records the subject's self-rated health on a vertical VAS with a score of 0-100, where the endpoints are labelled 0 for 'The worst health you can imagine' and 100 for 'The best health you can imagine'.
Time Frame: Through Week 14
Population: Full Analysis Set with all subjects with baseline and Week 14 data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 42 | 42
units on a scale | 2.9 (22.60) | 5.6 (15.28)

9. Secondary Outcome: Change From Baseline to Week 14 in Patient Global Impression of Change/Severity.
Description: The Patient Global Impression of Change (PGI-C) is a single question scale asking the patient to rate the overall status of their specific condition on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). The Patient Global Impression of Severity (PGI-S) is a single question scale asking the patient to rate current state of their specific condition on a 7-point scale ranging from 1 (normal) to 7 (extreme).
Time Frame: Through Week 14
Population: Full Analysis Set with all subjects with baseline and Week 14 data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 42 | 42
units on a scale
  PGI-S | 0.0 (1.28) | -0.4 (1.31)
  PGI-C | 3.4 (1.50) | 3.0 (1.63)

10. Secondary Outcome: Change From Baseline to Week 14 in Clinician Global Impression of Improvement/Severity.
Description: The Clinician Global Impression of Improvement (CGI-I) is a single question scale asking clinician to rate the overall status of the patient's specific condition on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). The Clinician Global Impression of Severity (CGI-S) is a single question scale asking the clinician to rate current state of the patient's specific condition on a 7-point scale ranging from 1 (normal) to 7 (extreme).
Time Frame: Through Week 14
Population: Full Analysis Set with all subjects with baseline and Week 14 data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 42 | 42
units on a scale
  CGI-S | -0.3 (0.86) | -0.5 (1.33)
  CGI-I | 3.4 (1.32) | 3.2 (1.52)

11. Secondary Outcome: The Number of Inhalations of Short-acting Beta Agonist (SABA) at Week 14.
Description: The number of times a short-acting beta agonist (number of inhalations) was used was assessed daily and reported as a weekly average.
Time Frame: Through Week 14
Population: Full Analysis Set with all subjects with baseline and Week 14 data available.
Measure: Mean (Standard Deviation); unit: number of inhalations
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 37 | 32
number of inhalations | 1.28 (1.507) | 0.97 (1.695)

12. Secondary Outcome: Change From Baseline to Week 14 in Serum Soluble LIGHT Levels (Lymphotoxin-like, Exhibits Inducible Expression, and Competes With Herpes Virus Glycoprotein D for Herpesvirus Entry Mediator, a Receptor Expressed by T Lymphocytes).
Description: Change from baseline in serum soluble LIGHT levels.
Time Frame: Through Week 14
Population: Full Analysis Set with all subjects with baseline and Week 14 data available.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 42 | 41
pg/mL | -114.52 (80.781) | 11.63 (92.147)

13. Secondary Outcome: Incidence of Anti-drug Antibodies (ADAs) at Each Timepoint.
Description: Incidence of anti-drug antibodies (ADAs) at Baseline, Week 2, Week 4, Week 6, Week 8, Week 12 and Week 14.
Time Frame: Baseline, Week 2, Week 4, Week 6, Week 8, Week 12 and Week 14.
Population: Safety Analysis Set: Data only collected for "AVTX-002" Arm/Group.
Measure: Count of Participants; unit: Participants
Arm/Group | AVTX-002 | Placebo
Number analyzed (Participants) | 45 | 0
Participants
  Baseline | 0 |
  Week 2 | 1 |
  Week 4 | 0 |
  Week 6 | 0 |
  Week 8 | 0 |
  Week 12 | 0 |
  Week 14 | 0 |

ADVERSE EVENTS:
Time Frame: Treatment emergent AEs were collected from the time of first dose through week 14 (14 weeks total).
Description: An AE will be considered treatment emergent if it occurs on or after the time (or date, if time not recorded) of first dose of IP and within 28 days after a subject's last dose of IP.
Arm/Group | AVTX-002 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 19/45 | 21/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVTX-002 (N=45) | Placebo (N=45)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT05288504/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/04/NCT05288504/SAP_001.pdf